CLINICAL TRIAL: NCT07241780
Title: The Effect of Live and Non-Living Parrot Therapy on Pain During Venous Blood Collection in Individuals With Chronic Diseases: A Double-Blind Randomized Controlled Study
Brief Title: Parrot Therapy on Pain During Venous Blood Collection in Individuals With Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Assistant professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RCS02072024
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pain; Chronic Disease
Keywords: Chronic disease; Pain management; Pet therapy; Venipuncture
MeSH Terms: conditions — Pain; Chronic Disease; Agnosia | interventions — Animal Assisted Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Live Parrot Group (Experimental): Before the venipuncture procedure began in the venipuncture unit, a nurse who was unaware of the details of the study (to prevent bias) administered the "Structured Patient Information Form" and "Visual Analogue Scale" to the patients. After the patient's venous blood was drawn by another nurse, the "Visual Analogue Scale " was administered again to measure the patients' pain levels during venipuncture.
  Interventions: Other: Live Parrot therapy (Pet therapy)
- Robotic Parrot Group (Experimental): Before the venipuncture procedure began in the venipuncture unit, a nurse who was unaware of the details of the study (to prevent bias) administered the "Structured Patient Information Form" and "Visual Analogue Scale" to the patients. After the patient's venous blood was drawn by another nurse, the "Visual Analogue Scale " was administered again to measure the patients' pain levels during venipuncture.
  Interventions: Other: Robotic Parrot therapy (Pet therapy)
- Picture Parrot Group (Experimental): Before the venipuncture procedure began in the venipuncture unit, a nurse who was unaware of the details of the study (to prevent bias) administered the "Structured Patient Information Form" and "Visual Analogue Scale" to the patients. After the patient's venous blood was drawn by another nurse, the "Visual Analogue Scale " was administered again to measure the patients' pain levels during venipuncture.
  Interventions: Other: Picture Parrot therapy (Pet therapy)
- Control Group (No Intervention): Before the venipuncture procedure began in the venipuncture unit, a nurse (to prevent bias) who was unaware of the study details administered the "Structured Patient Information Form" and the "Visual Analogue Scale" to the patients. After the patient's venous blood was collected by another nurse, the "Visual Analogue Scale" was administered again to measure the patients' pain levels during venipuncture. No other procedures were performed on these patients besides venipuncture.

INTERVENTIONS:
Other: Live Parrot therapy (Pet therapy) — During venipuncture, until the procedure was completed, patients interacted with a "Sultan parrot" (watching and talking) for approximately 5 minutes, depending on their group.
  Arms: Live Parrot Group
Other: Robotic Parrot therapy (Pet therapy) — During venipuncture, until the procedure was completed, patients interacted with a "robotic parrot" (watching and talking, listening to music) for approximately 5 minutes, depending on their group.
  Arms: Robotic Parrot Group
Other: Picture Parrot therapy (Pet therapy) — During venipuncture, until the procedure was completed, patients interacted with a "parrot picture" (examining and looking at pictures) for approximately 5 minutes, depending on their group.
  Arms: Picture Parrot Group

SUMMARY:
This double-blind randomized controlled trial was conducted to comparatively evaluate the effectiveness of live parrot, robotic parrot, and parrot picture therapies on pain during venipuncture in adults with chronic illness.

DETAILED DESCRIPTION:
Although venipuncture is a routine part of diagnostic and treatment processes, it is an invasive procedure that causes significant pain, anxiety, and physiological stress responses in individuals. This negative experience becomes a health problem, reduces treatment compliance, and can negatively affect quality of life, especially in individuals with chronic diseases such as diabetes and chronic kidney failure, who require regular follow-up and treatment. The systemic side effects and practical limitations of pharmacological pain control methods increase the need for safe, effective, and easy-to-apply non-pharmacological methods every day. In this context, distraction stands out as one of the most widely accepted mechanisms for modulating pain.

In the literature, the effect of non-pharmacological treatment methods reported to reduce pain and suffering is mostly explained by the gate control theory. According to the Gate Control Theory, the activity of thin and thick fibers located in the dorsal horn of the spinal cord acts as a gate that controls the sensation of pain. The activity of thin fibers opens this gate, while the activity of thick fibers closes it. When the gate is open, the pain signal reaches the conscious level, while when it is closed, the signal is prevented from reaching the conscious level. Therefore, by ensuring that patients receive intense stimulation through distraction methods such as pet therapy, the passage of pain signals to the brain stem is inhibited, and the patient's perception of pain is prevented.

In the pediatric population, parent-involved distraction and blowing a pinwheel, light-up toys, kaleidoscopes, blowing balloons, play dough, and watching cartoonshave been shown to significantly reduce pain. In adults, the Valsalva maneuver, the cough trick, music therapy, acupressure, and virtual reality have been reported to yield similarly positive results.

Animal-assisted therapies are gaining attention as a powerful non-pharmacological option in emotional and attentional contexts. In one study in children with type 1 diabetes found that interaction with a live animal was effective in reducing the pain of insulin injections. However, the use of live animals has significant limitations, such as infection control, allergy risk, animal welfare, the need for trained personnel, and cost. These limitations necessitate the exploration of alternative and more practical models. While robotic animals have the potential to overcome some of these challenges by offering realistic appearance and interaction, simple images can be considered a cost-free and universally applicable option. Parrots, in particular, are an attractive therapeutic tool in both live and robotic forms due to their colorful feathers, social nature, and mimicry skills. Indeed, the literature shows that even the use of animal-themed tubes or images can reduce pain and fear in children. However, no double-blind randomized controlled study has been found that directly compares the relative effectiveness of a live parrot, an advanced interactive robotic parrot, and a static parrot image in managing venipuncture pain in adults with chronic illness. This study was conducted to evaluate the effect of pet therapy (live parrot, robotic parrot, parrot image) applied using the three different attention-distraction methods mentioned above on venipuncture pain in individuals with chronic illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older,
* Literate,
* Able to communicate verbally,
* Without vision/hearing/speech problems,
* With at least 6 months of chronic disease,
* With a single venous access point, and who gave consent were included.

Exclusion Criteria:

* Refusal to give consent,
* Psychiatric diagnosis,
* Hemodynamic instability,
* Presence of Chronic Obstructive Pulmonary Disease/Asthma,
* Chronic disease duration of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Day 1
  The visual analogue scale is used to assess the intensity of pain experienced by individuals during acute pain. The scale consists of a vertical or horizontal line measuring 10 centimeter/100 millimeter in length, ranging from 0 points = no pain to 10 points = unbearable pain.
  In this project, it was used twice on each participant to determine their pain level before and during venipuncture.

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later